CLINICAL TRIAL: NCT00812123
Title: Open, Single Center, Randomised, Parallel Group Pilot Study to Investigate a Calcineurin Free Immunosuppressive Treatment for de Novo Renal Transplant Recipients: A Comparison of a Rapamycin/MMF/Steroids Regime to a Cyclosporine A Neoral/MMF/Steroids Regimen in the Prevention of Acute Rejection Following Renal Transplantation
Brief Title: Calcineurin Free Immunosuppression in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Prof. Dr. J. Steiger, University Hospital Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Calfree
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Kidney Transplantation; Chronic Kidney Disease
Keywords: kidney transplantation; calcineurin inhibitor free; protocol biopsy; Cyclosporin A; Sirolimus
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sirolimus; Cyclosporine; Prednisone; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcineurin free (Experimental): Immunosuppression with Sirolimus, Mycophenolate and Steroids
  Interventions: Drug: Sirolimus; Drug: Prednisone; Drug: Mycophenolate mofetil; Procedure: Protocol biopsies
- Calcineurin (Active Comparator): Immunosuppressive therapy with Cyclosporin A, Mycophenolate and Steroids
  Interventions: Drug: Cyclosporine A; Drug: Prednisone; Drug: Mycophenolate mofetil; Procedure: Protocol biopsies

INTERVENTIONS:
Drug: Sirolimus — Loading dose 30 mg for three days, trough level of 10-20 ng/ml month 1-3, 8-15 ng/ml month 4 - 6
  Other Names: Rapamune
  Arms: Calcineurin free
Drug: Cyclosporine A — Loading dose of 300 mg for three days, trough levels 250-300 ng/ml months 1-3, 150-250 ng/ml months 4 to 6
  Other Names: Sandimmun neoral
  Arms: Calcineurin
Drug: Prednisone — 0.5 mg/kg, tapering every two weeks until 0.1 mg/kg
Drug: Mycophenolate mofetil — 2 x 1000mg, through level above 2ug/ml
  Other Names: CellCept
Procedure: Protocol biopsies — protocol kidney biopsies at month one and three

SUMMARY:
The main purpose of this study is to obtain preliminary information on the efficacy, safety and cost of two regimens, Rapamycin / MMF / steroid therapy and Cyclosporine A Neoral / MMF / steroid therapy, used in the prevention of acute rejection following renal transplantation.

DETAILED DESCRIPTION:
This pilot study is designed to show differences in efficacy, safety and cost between the two regimens. Its main purpose is to provide information, if calcineurin free immunosuppressive treatment is a valuable alternative in the treatment of de novo kidney transplant recipients. Furthermore, by investigating the side effects in both arms it will be possible to decide, if the absence of calcineurin inhibition and lack of nephrotoxicity will outweigh the adverse effects of Rapamycin. With the obtained information it will be possible to plan a larger trial, which is warranted to compare the mentioned treatment regimens in more detail.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 15 and 75 years of age, regardless of race.
* Female patients of child bearing age agree to maintain effective birth control practice during the study.
* Patient has end stage kidney disease and is a suitable candidate for primary renal transplantation or retransplantation as assessed by the transplantation center.
* Patient has been fully informed and has given written or independent person witnessed oral informed consent.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient has a low immunological risk constellation, defined by receiving a kidney from a HLA-identical related living donor.
* Patient has a high immunological risk constellation, defined as having within the previous three years a measured PRA grade of ≥25% and/or having a previous graft survival shorter than 3 years due to rejection.
* Patient and donor have a positive T or B-cell crossmatch.
* Patient and donor are ABO incompatible.
* Age of donor > 68 years.
* Cold ischemia time > 36 hours.
* Patient has leucopenia, defined as having at transplantation less than 3000/mm3 leukocytes.
* Patient has thrombocytopenia, defined as having at transplantation less than 75000/mm3 thrombocytes.
* Patient is allergic or intolerant to cremophor RH 60 or structurally related compounds, steroids, Cyclosporine A Neoral, Rapamycin or MMF.
* Patient requires initial sequential or parallel therapy with immunosuppressive antibody preparation(s).
* Patient or donor is known to be HIV positive.
* Patient has significant liver disease, defined as having during the past 28 days continuously ASAT (SGOT) and/or ALAT (SGPT) levels greater than 3 fold of the upper value of the normal range of the investigational site.
* Patient with malignancy or history of malignancy ≥ 2 years, except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Patient has significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, or active peptic ulcer.
* Patient is taking or has been taking an investigational drug in the past 28 days.
* Patient has previously received or is receiving another organ transplant other than kidney.
* Patient is unlikely to comply with the visits schedule in the protocol.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2001-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Plasma Creatinine | 6 months

SECONDARY OUTCOMES:
Graft survival | 6 months
Patient survival | 6 months
Incidence of first acute rejections and number of total rejections | 6 months
Total number of anti-rejection treatments | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürg U Steiger, MD, Principal Investigator — Clinic for Transplantation Immunology and Nephrology, University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinic for Transplantation Immunology and Nephrology, Basel, Switzerland

REFERENCES:
- [Derived] Franz S, Regeniter A, Hopfer H, Mihatsch M, Dickenmann M. Tubular toxicity in sirolimus- and cyclosporine-based transplant immunosuppression strategies: an ancillary study from a randomized controlled trial. Am J Kidney Dis. 2010 Feb;55(2):335-43. doi: 10.1053/j.ajkd.2009.09.004. Epub 2009 Nov 17. PMID 19926370